CLINICAL TRIAL: NCT03138226
Title: Living Donor Uterus Transplantation Between Identical Twins
Acronym: UTx-twin
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: University Hospital Tuebingen (Other); University of Belgrade (Other)
Responsible Party: Principal Investigator, Mats Brännström, Professor, Sahlgrenska University Hospital
Other Study IDs: Twin UTx
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Absolute Uterine Factor Infertility; Cervical Cancer
Keywords: uterus, transplantation, infertility, twin
MeSH Terms: conditions — Uterine Cervical Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Cervical biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: uterus transplantation

SUMMARY:
Living donor uterus transplantation between identical twins, with IVF before and ET several months after transplantation. The donor should have completed childbirth.

DETAILED DESCRIPTION:
Living donor uterus transplantation between identical twins, with IVF before and ET several months after transplantation. The donor should have completed childbirth.

ELIGIBILITY:
Inclusion Criteria:

* age below 40 years
* absolute uterine factor infertility
* BMI<30-

Exclusion Criteria:

* systemic disease

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: absolute uterine factor infertility - monozygotic twin
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Live births after uterus transplantation | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Published in articles